CLINICAL TRIAL: NCT01668303
Title: Family-Based Juvenile Drug Court Services
Acronym: JDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Gayle Dakof, Associate Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA017478 (NIH)
Record Dates: First submitted 2012-08-06; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Substance Use; Delinquency
Keywords: juvenile drug court; adolescents; substance abuse; delinquency; family therapy; multidimensional family therapy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miami Juvenile Drug Court-MDFT (Experimental): Multidimensional family therapy (MDFT) is primarily a family-based approach (Liddle, 2002)which conducts individual sessions with the teen and parent[s] but not peer-group sessions.
  Interventions: Behavioral: Miami Juvenile Drug Court-MDFT
- Miami Juvenile Drug Court -TAU (Other): The Treatment as Usual (TAU) condition is primarily a peer group-based and individual approach that uses cognitive-behavioral principles and interventions.
  Interventions: Behavioral: Miami Juvenile Drug Court -TAU

INTERVENTIONS:
Behavioral: Miami Juvenile Drug Court-MDFT — MDFT assesses and intervenes in five domains: 1) Interventions with the adolescent, 2) interventions with the parent, 3) interventions to improve the parent-adolescent relationship, 4) interventions with other family members, and 5) interventions with external systems.
  Arms: Miami Juvenile Drug Court-MDFT
Behavioral: Miami Juvenile Drug Court -TAU — Each client is provided with a primary outpatient counselor who develops a treatment plan to address long-range goals. Family members are included in an assessment and treatment planning session at the beginning of treatment, but no formal family therapy is provided. Group therapy topics include self-esteem enhancement, decision-making skills, stress/anger management, communication skills, health education, teen pregnancy prevention, and occupational/career planning.
  Arms: Miami Juvenile Drug Court -TAU

SUMMARY:
The objective of the proposed study is to adapt and implement an efficacious adolescent substance abuse treatment, Multidimensional Family Therapy (MDFT), within the juvenile drug court service system. Additionally, the investigators will also examine the extent to which MDFT can enhance the effectiveness of existing juvenile drug court services in terms of decreasing drug use, delinquent behavior and arrests and improving school and vocational outcomes. The study design is a fully randomized controlled trial.

DETAILED DESCRIPTION:
Many questions remain regarding optimal treatments for juvenile drug court. To address this gap, the investigators will compare two treatments delivered in a drug court setting: Multidimensional Family Therapy (MDFT) and adolescent group therapy (AGT). This 5-year study will employ a fully randomized (2 conditions) by 5 assessment points (baseline, 6, 12, 18, and 24 months following baseline), repeated measures intent-to-treat design with multiple dependent variables. Adolescents who have been accepted into the Miami Juvenile Drug Court (MJDC) will be randomized to receive one of two treatments: MDFT (n = 57) or AGT (n = 55). The substance abuse treatments will be equivalent in terms of therapeutic dosage, and all youth with receive the same drug court program with wtreatment received being the only difference (family vs non-family treatment). In order to maximize the ecological validity of the study, both treatments will be delivered by community-based drug abuse counselors. MDFT will be delivered by providers at Jackson Memorial Hospital's Adolescent Substance Abuse Program and AGT by providers at a separate facility, Here's Help.

Aim 1. Acceptability and Effectiveness. The study will address the comparative acceptability and effectiveness of the two drug court programs in ways that are consistent with recommendations from the juvenile drug court literature to consider multi-domain and multiple perspectives of program goals and outcomes. First, effectiveness will be assessed in terms of the differential rates at which youth in MDFT and AGT graduate from drug court, a primary goal of the drug court program. Juvenile offending substance abusers and their families are notoriously difficult to engage and retain in any type of treatment program, yet family-based interventions have demonstrated impressive retention rates with these populations. Thus an important aspect of the proposed effectiveness evaluation will be the extent to which the MDFT intervention improves drug court program completion rates. Our second perspective on effectiveness involves an examination of the rates of change in a number of critical domains, including reductions in substance use, arrests, and delinquent behaviors, as well as improvements in school/vocational performance over a 2-year period. With these multidimensional outcome assessments the investigators will be able to explore different dimensions and trajectories of recovery following drug court participation. This is consistent with the aims of juvenile drug courts not only to reduce drug use and delinquency but also to increase adolescents' prosocial skills and behaviors. The investigators are also interested in examining multiple perspectives on the relative acceptability of MDFT to drug court staff, teens, and families, as recommended by drug court researchers.

Aim 2. Drug Court Program Mechanisms. While the few existing studies of key drug court factors have focused mainly on the structural and judicial aspects of drug court programs, almost nothing is known about the treatment processes affecting drug court outcomes, or the mechanisms of clinical and judicial component impact. Clearly, an important next step in this specialty is to delineate the treatment processes and ingredients that maximize outcomes in drug court, particularly in relation to the application of evidence-based therapy models within drug court programs. Examination of change mechanisms is now recognized as an essential feature of state-of-the-art drug abuse intervention research. Among those process variables considered important in mediating drug treatment outcomes are the therapeutic alliance that is formed between provider and client , and the extent to which a positive collaborative relationship develops among all drug court team members, including the judge. Research on family-based interventions supports the contention that family-based treatments exert their effects through the reduction of family risk and the facilitation of protective processes, and family functioning has been found to play a primary role in helping teens achieve and maintain recovery after substance abuse treatment. In sum, given that the quest to improve drug court program development, implementation, and outcomes rests in large part on the clarification of the programs' mechanisms of action, drug court researchers have turned their attention to analyses linking within-program processes to outcomes. The proposed study will do likewise.

ELIGIBILITY:
Inclusion Criteria:

(a) Substance abuse or dependence disorder requiring outpatient treatment, and (b)after consulting with his or her attorney, the youth and family voluntarily agrees to enter juvenile drug court.

Exclusion Criteria:

(a) Their current offense is the sale of drugs, a gun offense, a violent offense, or sexual battery,(b) their current offense is likely to merit commitment to a secure or locked juvenile justice facility or (c) they have severe mental illness or retardation according to their intake MJDC evaluation.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2004-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Graduation from juvenile drug court | Collected once at 12 months from intake/baseline.
  Status of drug court graduation (graduated from drug court or did not graduate from drug court)
Change in substance use | Baseline at the begining of the study, and then at 6, 12, 18, and 24 months after baseline
  Personal Experiences with Chemicals Inventory
Change in delinquency | Baseline, and then at 6, 12, 18, and 24 months after baseline
  Self-report, parent report, and juvenile justice records: Self-report delinquency scale, Youth Self Report, Child Behavior Checklist; arrests and disposition from juvenile justice records.
Change in Mental health symptoms | Baseline, 6, 12, 18 and 24 months after baseline
  Youth and parent report: Child Behavior Checklist, Youth Self Report
Change in Family functioning | Baseline, 6, 14, 18, and 24 months after baseline
  Youth and Parent Report: Family Environment Scales, Parental Stress Index, Behavior Affect Relationship Scales
Length of treatment | Collected once, at 12 months after baseline
  How many weeks of treatment received
Change in arrests | 12 months before intake through 24 months after intake
  Arrests will be extracted from juvenile justice records.
Change in substance use | Intake, 6, 12, 18, 24 months after intake
  Measured by the Timeline Follow Back Method
Change in substance use | Intake, 6, 12, 18 and 24 months after intake
  Urinanalysis to detect drugs

CONTACTS AND LOCATIONS:
Overall Officials: Gayle A. Dakof, Ph.D., Principal Investigator — University of Miami
Locations (4):
- United States (4):
  - Here's Help Inc., Miami, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Juvenile Drug Court, Miami, Florida

REFERENCES:
- [Derived] Dakof GA, Henderson CE, Rowe CL, Boustani M, Greenbaum PE, Wang W, Hawes S, Linares C, Liddle HA. A randomized clinical trial of family therapy in juvenile drug court. J Fam Psychol. 2015 Apr;29(2):232-41. doi: 10.1037/fam0000053. Epub 2015 Jan 26. PMID 25621927